CLINICAL TRIAL: NCT01820819
Title: Is Access to Liver Transplantation Similar in Alcoholic or Not Patients? A Prospective Cohort Study
Brief Title: Is Access to Liver Transplantation Similar in Alcoholic or Not Patients?
Acronym: TRANSALC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Saint Antoine Hospital (Pr Yvon Camus) (Unknown)
Responsible Party: Sponsor
Other Study IDs: AOM 10003
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Inpatient With End Stage Liver Disease
Keywords: Inpatient; Liver cirrhosis; Liver Cirrhosis, Alcoholic; Physician's Practice Patterns; Liver Transplantation; Delivery of Health Care; Resource Allocation
MeSH Terms: conditions — Liver Cirrhosis; Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Registered or not on the transplantation national waiting list

SUMMARY:
The purpose of this study is to determine whether there are reasons other than medical reasons that could limit access to liver transplantation in alcoholic patients.

DETAILED DESCRIPTION:
The investigators perform a study combining the follow up of a previous cohort of 450 patients and the inclusion of 150 new patients.

The study is performed in medical or hepatogastroenterology departments of nine French public hospitals mostly non-teaching. They lay in three French area, selected according to the density of patients with alcoholic liver disease (ALD) in the area, respectively, "high" as in Brittany-Loire, 'average' in Ile de France and "low" as in the Languedoc-Roussillon.

The patients included in the cohort must respond to the following criteria: having liver cirrhosis of whatever origin and age over 18 years. The cirrhosis must be confirmed by the morphological or histological criteria.

Structured forms and questionnaires will allow the collection of data. Information collected from patients include socio demographic characteristics, medical history, history of consumption of psychotropic (i.e., alcohol or drugs), clinical, biological, histological characteristics and psychological. Inpatients complete a self-assessment structured questionnaire "Hospital Anxiety Depression Scale" (HAD).

Patients are followed until they are registered or not on the national waiting list or die, every 6 months after inclusion until 2 years.

Statistical analysis will focus on descriptive analysis, survival analysis by Kaplan-Meier, and analytic analysis. Association with registration on the national waiting list of inpatients will be searched using Cox and logistic regression models. Further analyzes will be conducted for example on the differences of opinion between physicians and patients, on regional differences.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* Age over 18
* Having liver cirrhosis of whatever origin (Cirrhosis was confirmed if morphological or histological criteria with or without esophageal varicoses were met)

Exclusion Criteria:

* Outpatients
* Age less to 18
* With acute liver failure or hepatocarcinoma without liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients aged over 18 admitted to medical or hepato gastroenterology departments of the hospitals selected in three French area with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 574 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Registration on the national waiting list | 3 years

SECONDARY OUTCOMES:
Potential candidate to liver transplantation according to the opinion of the caring physician on | At Day 0
  At the time of inpatients inclusion (previous study: fifth year after the first inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Yvon Calmus, MD, PhD, Study Director — Paris-Est University, AP-HP
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Background] Perut V, Conti F, Scatton O, Soubrane O, Calmus Y, Vidal-Trecan G. Might physicians be restricting access to liver transplantation for patients with alcoholic liver disease? J Hepatol. 2009 Oct;51(4):707-14. doi: 10.1016/j.jhep.2009.04.018. Epub 2009 May 28. PMID 19665248
- [Background] Cohen C, Benjamin M. Alcoholics and liver transplantation. The Ethics and Social Impact Committee of the Transplant and Health Policy Center. JAMA. 1991 Mar 13;265(10):1299-301. doi: 10.1001/jama.265.10.1299. PMID 1995978
- [Background] Lucey MR, Beresford TP. Alcoholic liver disease: to transplant or not to transplant? Alcohol Alcohol. 1992 Mar;27(2):103-8. PMID 1524600
- [Background] Ubel PA. Transplantation in alcoholics: separating prognosis and responsibility from social biases. Liver Transpl Surg. 1997 May;3(3):343-6. PMID 9346761
- [Result] Vidal-Trecan G, Kone V, Pilette C, Nousbaum JB, Doll J, Buffet C, Eugene C, Podevin P, Boutet O, Puyeo J, Conti F, Calmus Y. Subjective parameters markedly limit the referral of transplantation candidates to liver transplant centres. Liver Int. 2016 Apr;36(4):555-62. doi: 10.1111/liv.13030. Epub 2015 Dec 21. PMID 26604165